CLINICAL TRIAL: NCT04200690
Title: Effectiveness of Interdisciplinary Combined Dermatology-Gastroenterology-Rheumatology Clinical Care Compared to Usual Care in Patients With Immune-Mediated Inflammatory Diseases: A Parallel Group, Non-blinded, Pragmatic Randomized Trial
Brief Title: Effectiveness of Interdisciplinary Care Compared to Usual Care in Patients With Immune-Mediated Inflammatory Diseases
Acronym: NCAS-1
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: NCAS-1
Record Dates: First submitted 2019-12-10; First posted 2019-12-16 (Actual); Last update posted 2023-06-02 (Actual); Status verified 2023-05

CONDITIONS: Psoriasis; Psoriatic Arthritis; Axial Spondyloarthritis; Hidradenitis Suppurativa; Crohn Disease; Ulcerative Colitis
MeSH Terms: conditions — Psoriasis; Arthritis, Psoriatic; Axial Spondyloarthritis; Hidradenitis Suppurativa; Crohn Disease; Colitis, Ulcerative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interdisciplinary management (Experimental): Interdisciplinary combined clinical care
  Interventions: Other: Interdisciplinary management
- Usual-care management (Active Comparator): Usual-care
  Interventions: Other: Usual-care management

INTERVENTIONS:
Other: Interdisciplinary management — The intervention in this trial consists of the combined efforts of the interdisciplinary team in the combined clinic arm.
  The interdisciplinary team consists of dermatologists, gastroenterologists, rheumatologists, nurses, psychologists, dieticians, social workers, physiotherapists, and secretaries. Treatment will be individualized based on clinical, biomarker, phenotypic, and psychosocial characteristics. The medical treatment will follow local, national and international guidelines.
  Arms: Interdisciplinary management
Other: Usual-care management — Usual care will be carried out by HCPs that are not otherwise involved in the trial. In usual care the patients will not be offered an interdisciplinary patient-centered care as described, but only attend their usual disease-specific departments at the usual appointments.Treatment will be prescribed as felt appropriate according to local, national and international guidelines by the treating physicians with no set protocol and no restrictions.
  Arms: Usual-care management

SUMMARY:
The overall aim of this study is to determine the effectiveness of an interdisciplinary combined clinic intervention compared to usual care in a population of patients with two or more Immune-mediated inflammatory diseases (IMIDs).

DETAILED DESCRIPTION:
Immune-mediated inflammatory diseases (IMIDs) such as psoriasis, hidradenitis suppurative, spondyloarthritis, and inflammatory bowel disease, are associated with increased risk of somatic and psychiatric comorbidities as well as reduced socioeconomic status and a risk of further autoimmune diseases. The unmet needs in the care of patients with IMIDs are caused by a lack of patient-centricity in the usual specialized siloed approach to these diseases. The overall aim of this study is to determine the effectiveness of an interdisciplinary combined clinic intervention compared to usual care in a population of patients with the IMIDs: psoriasis, hidradenitis suppurativa, spondyloarthritis, ulcerative colitis, and Crohn's disease. This trial is designed to determine if the interdisciplinary intervention works in a real-world setting and thus has several pragmatic elements. The hypotheses will be tested in a randomized, usual care controlled, parallel-group clinical trial. Consecutively enrolled subjects are randomly assigned in a 2:1 ratio to either treatment in the interdisciplinary combined clinic or usual care in a hospital clinical setting. 300 subjects (anticipated) will be randomized to either multidisciplinary combined clinic intervention (200 subjects, anticipated) or usual care (100 subjects, anticipated). The study will consist of a 24-Week active intervention period and an additional 24-Weeks follow-up period.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent obtained from the subject prior to randomization.
2. Age 18 and above.
3. Diagnosis of at least two IMIDs* or diagnosis of one IMID and clinical suspicion** of another IMID*

   * including and limited to: Psoriasis, HS, UC, CD, axSpA, PsA ** substantiated by e.g. clinical findings, imaging, biochemical results or histological examination at the discretion of the investigator.

Exclusion Criteria:

1. Non-Danish speaking
2. Expected to be unable to comply with the study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2020-01-14 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2024-01-31 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline on the Short-Form Health Survey (SF-36) Physical Component Summary (PCS) | 24 Weeks
  SF-36 is a patient-reported outcome (PRO) measure evaluating a participant's health status. It comprises 36 items covering 8 domains: physical functioning, role physical, role emotional, bodily pain, vitality, social functioning, mental health, and general health. Items are answered on Likert scales of varying lengths. Items from 8 domains contribute to the PCS. The summary scores range from 0 to 100, with higher scores indicating better levels of function and/or better health.
Change From Baseline on the Short-Form Health Survey (SF-36) Mental Component Summary (MCS) | 24 Weeks
  SF-36 is a patient-reported outcome measure evaluating a participant's health status. It comprises 36 items covering 8 domains: physical functioning, role physical, role emotional, bodily pain, vitality, social functioning, mental health, and general health. Items are answered on Likert scales of varying lengths. Items from 8 domains contribute to the MCS. The summary scores range from 0 to 100, with higher scores indicating better levels of function and/or better health.

SECONDARY OUTCOMES:
Proportion of subjects achieving Minimal Clinical Important Difference (MCID) on the Short-Form Health Survey (SF-36) Physical Component Summary (PCS) | 24 Weeks
  SF-36 is a patient-reported outcome (PRO) measure evaluating a participant's health status. It comprises 36 items covering 8 domains: physical functioning, role physical, role emotional, bodily pain, vitality, social functioning, mental health, and general health. Items are answered on Likert scales of varying lengths. Items from 8 domains contribute to the PCS. The summary scores range from 0 to 100, with higher scores indicating better levels of function and/or better health.
Change From Baseline in the Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-Fatigue) Score | Week 24
  The FACIT-Fatigue scale is a 13-item self-administered questionnaire that assesses both the physical and functional consequences of fatigue. Each question is answered on a 5-point scale, where 0 means "not at all," and 4 means "very much." The FACIT-Fatigue scale score ranges from 0 to 52, with higher scores denoting lower levels of fatigue. A positive change from Baseline score indicates an improvement.
Change from baseline in the Work Productivity and Activity Impairment Questionnaire (WPAI:GH) Percentage of Overall Work Impairment | Week 24
  The WPAI assess the impact of disease on work productivity and daily activities during the past seven days, using 6 questions regarding: 1 (if currently employed); 2 (hours missed due to disease); 3 (hours missed other reasons); 4 (hours actually worked); 5 (degree disease affected productivity while working); 6 (degree disease affected regular activities). WPAI generates four main outcomes: 1 percentage of work time missed (absenteeism); percentage of impairment while working (presentisms); percentage of overall work impairment (absenteeism and presentisms combined); and percentage of activity impairment. Scores for WPAI range from 0% to 100%, where 0 % indicates no impairment and 100% is total loss of work productivity/activity.
Change in mean General Self-Efficacy scale scores | Week 24
  The General Self-Efficacy Scale is a 10-item psychometric scale that is designed to assess optimistic self-beliefs to cope with a variety of difficult demands in life.
Change in the mean Hospital Anxiety and Depression Scale - Anxiety (HADS-A) | Week 24
  14-item measure designed to assess anxiety and depression symptoms in medical patients, with emphasis on reducing the impact of physical illness on the total score. The depression items tend to focus on the anhedonic symptoms of depression. Items are rated on a 4-point severity scale. The HADS produces two scales, one for anxiety (HADS-A) and one for depression (HADS-D), differentiating the two states.
Change in the mean Hospital Anxiety and Depression Scale - Anxiety (HADS-D) | Week 24
  14-item measure designed to assess anxiety and depression symptoms in medical patients, with emphasis on reducing the impact of physical illness on the total score. The depression items tend to focus on the anhedonic symptoms of depression. Items are rated on a 4-point severity scale. The HADS produces two scales, one for anxiety (HADS-A) and one for depression (HADS-D), differentiating the two states.

OTHER OUTCOMES:
Change From Baseline in Dermatology Life Quality Index (DLQI) | 24 and 48 Weeks
  The DLQI is a 10-item questionnaire that measures the impact of skin disease on participant's quality of life. Each question was evaluated on a 4-point scale ranging from 0 (not at all) to 3 (very much); where higher scores indicate more impact on quality of life. The DLQI total score ranges from 0 (not at all) to 30 (very much). Higher scores indicate more impact on quality of life of participants.
Change From Baseline in Health Assessment Questionnaire- Disability Index (HAQ-DI) | 24 and 48 Weeks
  The Health Assessment Questionnaire - Disability Index is a patient-reported questionnaire consisting of 20 questions referring to eight domains: dressing/grooming, arising, eating, walking, hygiene, reach, grip, and usual activities. Participants assessed their ability to do each task over the past week using the following response categories: without any difficulty (0); with some difficulty (1); with much difficulty (2); and unable to do (3). Scores on each task are summed and averaged to provide an overall score ranging from 0 to 3, where zero represents no disability and three very severe, high-dependency disability. Negative mean changes from Baseline in the overall score indicate improvement in functional ability.
Change in the mean Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) | 24 and 48 Weeks
  The BASDAI is used for measuring and evaluating disease activity in ankylosing spondylitis. This index consists of 6 questions pertaining to the 5 major symptoms of ankylosing spondylitis: fatigue, spinal pain, joint pain/swelling, areas of localized tenderness (or enthesitis, defined as inflammation of tendons and ligaments), duration of morning stiffness, severity of morning stiffness. A visual analogue scale ranging from 0 (none) to 10 (very severe) is used to answer the questions. The final BASDAI score averages the individual assessments for a final score range of 0 to 10 (0 being no problem and 10 being the worst problem).
Change from baseline in the Short Inflammatory Bowel Disease Questionnaire (SIBDQ) Total Score | 24 and 48 Weeks
  The SIBDQ is a disease-specific health-related quality of life (HRQoL) questionnaire, able to detect and define meaningful clinical changes in inflammatory bowel disease (IBD) patients by measuring physical, social and emotional status. The SIBDQ consists of 10 questions, each question is scored on a scale from 1 (poor QoL) to 7 (good QoL). The scores are summed up and range from 10 (poor QoL) to 70 (good QoL). A higher score indicates a better HRQoL; a positive change from baseline indicates improvement.
Change from baseline in body weight | 24 and 48 Weeks
  Change in body weight (kg)
Change from baseline in blood lipid levels | 24 Weeks
  Lipid panel included low density lipoprotein (LDL) cholesterol, high density lipoprotein (HDL) cholesterol, total cholesterol, and triglycerides.
Improvement in Psoriasis Area and Severity Index (PASI) | 24 Weeks
  The PASI is a system used for assessing and grading the severity of psoriatic lesions. In the PASI system, the body is divided into 4 regions: the head, trunk, upper extremities, and lower extremities. Each of these area was assessed separately for the percentage of the area involved, which translates to a numeric score that ranges from 0 to 6, and for erythema, induration, and scaling, which are each rated on a scale of 0 to 4. The PASI produces a numeric score that can range from 0 to 72. A higher score indicates more severe disease.
The proportion of participants who achieve ASDAS remission (remission <1.3 / not in ASDAS remission >1.3) based on the Ankylosing Spondylitis Disease Activity Score (ASDAS) measure | 24 Weeks
  ASDAS remission is a score of <1.3 on a composite index to assess disease activity in Ankylosing Spondylitis. Parameters include spinal pain, the patient's global assessment of disease activity, peripheral pain/swelling, duration of morning stiffness and C-reactive protein (CRP) in mg/L.
The proportion of participants who achieve an ASAS 20 / 40 response (Assessment of SpondyloArthritis International Society criteria) | 24 Weeks
  ASAS 20 / 40 response is a validated composite assessment, reflecting the proportion of treated patients who achieve within a defined time frame at least 20% / 40% improvement in score in at least 3 of a conventional set of 4 clinical domains relevant to AS and no worsening in the fourth domain.
Percentage of Participants With an ACR 20/40 Response | 24 Weeks
  Percentage of participants with an American College of Rheumatology 20% / 40% (ACR20/40) response at Week 24. A participant is a responder if the following 3 criteria for improvement from Baseline are met: • ≥ 20% / 40% improvement in 68 tender joint count; ≥ 20% / 40% improvement in 66 swollen joint count; and ≥ 20% improvement in at least 3 of the 5 following parameters: Patient's assessment of pain (measured on a 100 mm visual analog scale [VAS]); Patient's global assessment of disease activity (measured on a 100 mm VAS); Physician's global assessment of disease activity (measured on a 100 mm VAS); Patient's self-assessment of physical function (Health Assessment Questionnaire - Disability Index (HAQ-DI)); C-Reactive Protein.
Percentage of patients achieving clinical response based on Harvey-Bradshaw Index (HBI) | 24 Weeks
  Clinical response is defined as a decrease in HBI score of >=3 points from baseline. HBI score is used to measure the disease activity of CD. It consists of clinical parameters: general well-being (0-4, where higher score means lower well being), abdominal pain (0-3, higher score means more severe pain), number of liquid stools per day, abdominal mass (0-3, where higher score means presence of swelling in the abdomen), and complications (score 1 per item). Total score is the sum of individual parameters. The score ranges from a minimum score of 0 to no pre-specified maximum score as it depends on the number of liquid stools, where higher scores indicating more severe disease.
Percentage of Participants achieving a clinical response <=2 based on the Simple Clinical Colitis Activity Index (SCCAI) | 24 Weeks
  The SCCAI measures disease activity as defined by both participants and examiners and includes the following 13 items: general well-being, abdominal pain, bowel frequency, stool consistency, bleeding, anorexia, nausea or vomiting, abdominal tenderness, extra-intestinal complications (eye, mouth, joint, skin), temperature, sigmoidoscopic assessment, nocturnal bowel movements, and urgency of defecation. Scores range from 0 to 19 points.
Proportion of patients with Hidradenitis Suppurativa Clinical Response (HiSCR) | 24 Weeks
  HiSCR is defined as at least a 50% decrease in Abscess and Inflammatory Nodule (AN) count with no increase in the number of abscesses or in the number of draining fistulae.
Change From Baseline on the Short-Form Health Survey (SF-36) Physical Component Summary (PCS) | 48 Weeks
  SF-36 is a patient-reported outcome (PRO) measure evaluating a participant's health status. It comprises 36 items covering 8 domains: physical functioning, role physical, role emotional, bodily pain, vitality, social functioning, mental health, and general health. Items are answered on Likert scales of varying lengths. Items from 8 domains contribute to the PCS. The summary scores range from 0 to 100, with higher scores indicating better levels of function and/or better health.
Change From Baseline on the Short-Form Health Survey (SF-36) Mental Component Summary (MCS) | 48 Weeks
  SF-36 is a patient-reported outcome measure evaluating a participant's health status. It comprises 36 items covering 8 domains: physical functioning, role physical, role emotional, bodily pain, vitality, social functioning, mental health, and general health. Items are answered on Likert scales of varying lengths. Items from 8 domains contribute to the MCS. The summary scores range from 0 to 100, with higher scores indicating better levels of function and/or better health.
Change in mean General Self-Efficacy scale scores | 48 Weeks
  The General Self-Efficacy Scale is a 10-item psychometric scale that is designed to assess optimistic self-beliefs to cope with a variety of difficult demands in life.
Change in the mean Hospital Anxiety and Depression Scale - Anxiety (HADS-D) | 48 Weeks
  14-item measure designed to assess anxiety and depression symptoms in medical patients, with emphasis on reducing the impact of physical illness on the total score. The depression items tend to focus on the anhedonic symptoms of depression. Items are rated on a 4-point severity scale. The HADS produces two scales, one for anxiety (HADS-A) and one for depression (HADS-D), differentiating the two states.
Change in the mean Hospital Anxiety and Depression Scale - Anxiety (HADS-A) | 48 Weeks
  14-item measure designed to assess anxiety and depression symptoms in medical patients, with emphasis on reducing the impact of physical illness on the total score. The depression items tend to focus on the anhedonic symptoms of depression. Items are rated on a 4-point severity scale. The HADS produces two scales, one for anxiety (HADS-A) and one for depression (HADS-D), differentiating the two states.
Change from baseline in the Work Productivity and Activity Impairment Questionnaire (WPAI:GH) Percentage of Overall Work Impairment | 48 Weeks
  The WPAI assess the impact of disease on work productivity and daily activities during the past seven days, using 6 questions regarding: 1 (if currently employed); 2 (hours missed due to disease); 3 (hours missed other reasons); 4 (hours actually worked); 5 (degree disease affected productivity while working); 6 (degree disease affected regular activities). WPAI generates four main outcomes: 1 percentage of work time missed (absenteeism); percentage of impairment while working (presentisms); percentage of overall work impairment (absenteeism and presentisms combined); and percentage of activity impairment. Scores for WPAI range from 0% to 100%, where 0 % indicates no impairment and 100% is total loss of work productivity/activity.
Change From Baseline in the Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-Fatigue) Score | 48 Weeks
  The FACIT-Fatigue scale is a 13-item self-administered questionnaire that assesses both the physical and functional consequences of fatigue. Each question is answered on a 5-point scale, where 0 means "not at all," and 4 means "very much." The FACIT-Fatigue scale score ranges from 0 to 52, with higher scores denoting lower levels of fatigue. A positive change from Baseline score indicates an improvement.

CONTACTS AND LOCATIONS:
Overall Officials: Kasper F Hjuler, MD PhD, Principal Investigator — Aarhus University Hospital; Lars Iversen, MD PhD DMSc, Study Chair — University of Aarhus
Locations (1):
- National Center for Autoimmune Diseases, Aarhus University Hospital, Aarhus, Denmark

REFERENCES:
- [Derived] Hjuler KF, Dige A, Agnholt J, Laurberg TB, Loft AG, Moller LF, Christensen R, Iversen L. Effectiveness of interdisciplinary combined dermatology-gastroenterology-rheumatology clinical care compared to usual care in patients with immune-mediated inflammatory diseases: a parallel group, non-blinded, pragmatic randomised trial. BMJ Open. 2021 Apr 28;11(4):e041871. doi: 10.1136/bmjopen-2020-041871. PMID 33910945